CLINICAL TRIAL: NCT03797469
Title: Nutritional Supplements and Performance During Visual Field Testing
Brief Title: Nutritional Supplements and Performance During Visual Field Testing (B3 Vitamin)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey Liebmann, Professor of Ophthalmology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AAAR8208
Record Dates: First submitted 2018-05-28; First posted 2019-01-09 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Visual Field Defect, Peripheral; Glaucoma, Open-Angle
Keywords: Perimetry; Vitamins; Glaucoma; Supplements; Vitamin B3; Nicotinamide
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Niacinamide; Pyruvic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide and Pyruvate (N&P) (Active Comparator): This group will receive two separate sets of tablets containing 3 x 1000 mg of Vitamin B3 (nicotinamide) and 2 x 1500 mg of Pyruvate.
  Interventions: Dietary Supplement: Vitamin B3; Dietary Supplement: Pyruvate
- Placebo (Placebo Comparator): This group will receive an equal number of tablets as the N&P group.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B3 — 3 tablets of 1000 mg each will be administered orally.
  Other Names: B-3 Nicotinamide
  Arms: Nicotinamide and Pyruvate (N&P)
Dietary Supplement: Pyruvate — 2 tablets of 1500 mg each will be administered orally.
  Other Names: Calcium Pyruvate
  Arms: Nicotinamide and Pyruvate (N&P)
Dietary Supplement: Placebo — Tablets will look identical to the supplements and the number of tablets will equal the amount of supplements provided.
  Arms: Placebo

SUMMARY:
This study seeks to test whether these over-the-counter nutritional supplements have an impact on patients' performance during visual field testing.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide. The most important test to detect progression is visual field testing. Visual field testing is the reference standard to measure visual function in glaucoma. It is called called standard automated perimetry (SAP). However, this test is very subjective, often unreliable, and variable. One of the main causes of unreliable tests is the lack of attentiveness or concentration during the test. Previous studies have shown that listening to Mozart or taking vitamin B12 can improve the reliability of this test. Recent studies have suggested that over-the-counter medications such as nicotinamide (vitamin B3) and pyruvate can also improve the performance during this test. This can ultimately reduce costs due to repeated testing and increase doctor's certainty when analyzing the results of this test.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary open-angle glaucoma;
* Visual field loss on 24-2 standard automated perimetry (SAP) worse than -3 decibels (dB) and better than -12 dB in both eyes;
* Best corrected visual acuity better than 20/40 in both eyes;
* Prior experience with 24-2 visual fields (at least 3 tests done in the past 3 years).

Exclusion Criteria:

* Significant cataract or media opacity;
* Diagnosis of dementia, Alzheimer's, and other neurological diseases;
* Current use or use in the past 1 month of nutritional supplements;
* Inability to take or intolerance to nicotinamide and/or pyruvate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 24-2 visual field test | Up to 20 weeks
  Changes in 24-2 visual field results based upon point-wise and global metrics before and after intervention, and between treatment and placebo groups will be compared.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) scores | Up to 20 weeks
  Montreal Cognitive Assessment (MoCA) score before and after intervention and correlate these changes with those seen on visual field tests will be compared. The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that assesses different types of cognitive abilities. Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Liebmann, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams PA, Harder JM, Cardozo BH, Foxworth NE, John SWM. Nicotinamide treatment robustly protects from inherited mouse glaucoma. Commun Integr Biol. 2018 Jan 19;11(1):e1356956. doi: 10.1080/19420889.2017.1356956. eCollection 2018. PMID 29497468
- [Background] Zhang M, Ying W. NAD+ Deficiency Is a Common Central Pathological Factor of a Number of Diseases and Aging: Mechanisms and Therapeutic Implications. Antioxid Redox Signal. 2019 Feb 20;30(6):890-905. doi: 10.1089/ars.2017.7445. Epub 2018 Feb 7. PMID 29295624
- [Background] Williams PA, Harder JM, John SWM. Glaucoma as a Metabolic Optic Neuropathy: Making the Case for Nicotinamide Treatment in Glaucoma. J Glaucoma. 2017 Dec;26(12):1161-1168. doi: 10.1097/IJG.0000000000000767. PMID 28858158
- [Background] Liebmann JM, Cioffi GA. Nicking Glaucoma with Nicotinamide? N Engl J Med. 2017 May 25;376(21):2079-2081. doi: 10.1056/NEJMcibr1702486. No abstract available. PMID 28538117
- [Background] Williams PA, Harder JM, Foxworth NE, Cardozo BH, Cochran KE, John SWM. Nicotinamide and WLDS Act Together to Prevent Neurodegeneration in Glaucoma. Front Neurosci. 2017 Apr 25;11:232. doi: 10.3389/fnins.2017.00232. eCollection 2017. PMID 28487632
- [Background] Williams PA, Harder JM, Foxworth NE, Cochran KE, Philip VM, Porciatti V, Smithies O, John SW. Vitamin B3 modulates mitochondrial vulnerability and prevents glaucoma in aged mice. Science. 2017 Feb 17;355(6326):756-760. doi: 10.1126/science.aal0092. PMID 28209901
- [Derived] De Moraes CG, John SWM, Williams PA, Blumberg DM, Cioffi GA, Liebmann JM. Nicotinamide and Pyruvate for Neuroenhancement in Open-Angle Glaucoma: A Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2022 Jan 1;140(1):11-18. doi: 10.1001/jamaophthalmol.2021.4576. PMID 34792559